CLINICAL TRIAL: NCT03236402
Title: "A Cross-sectional Comparative Study to Assess Knowledge and Opinion Regarding Adoption Among Adults Residing in Rural and Urban Area of Ambala, Haryana"
Brief Title: "A Study to Assess Knowledge and Opinion Regarding Adoption Among Adults Residing in Rural and Urban Area"
Status: Completed | Type: Observational
Sponsor: Maharishi Markendeswar University (Deemed to be University) (Other)
Responsible Party: Principal Investigator, Santosh Kumari, Principal Investigator, Maharishi Markendeswar University (Deemed to be University)
Other Study IDs: 100015
Record Dates: First submitted 2017-07-19; First posted 2017-08-01 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Knowledge
Keywords: Knowledge; Opinion; Adoption; Adults; Cross-Sectional

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Early young adult (20 years - 30 years): Adults who were in the age group of 20 - 30 years was the first group. There were made two separate same age group one for rural and one for urban areas adults. Each areas age group consist 50 adults of 20-30 years.
- Middle age adult (31 -50 years): Adults who were in the age group of 31-50 years were in second group. There were made two separate same age group one for rural and one for urban areas adults. Each areas age group consist 50 adults of 31-50 years.
- Late adult (51 years - 65 years): Adults who were in the age group of 51-65 years were in third group. There were made two separate same age group one for rural and one for urban areas adults. Each areas age group consist 50 adults of 51-65 years.
- >65 years: Adults who were in the age group of >65 years were in fourth group. There were made two separate same age group one for rural and one for urban areas adults. Each areas age group consist 50 adults of >65 years.

SUMMARY:
A cross - sectional comparative study to assess knowledge and opinion regarding adoption among adults residing in rural and urban area of Ambala, Haryana.

DETAILED DESCRIPTION:
ABSTRACT INTRODUCTION: Children are regarded as the precious gift in world. It is estimated that between 8% and 12% of couples worldwide suffer from infertility with rate of 10% in India and about 20 million children are orphan even then adoption rates are falling in India.

OBJECTIVES: To assess and compare the knowledge score and opinion score regarding adoption among adults of different age groups.To determine relationship between knowledge and opinion regarding adoption among adults.To seek association of knowledge score and opinion score regarding adoption with selected variables.

METHODOLOGY: A descriptive cross sectional survey design was used. 400 adults of rural (200) and urban (200) area were selected by using quota sampling technique. The data was collected by structured knowledge questionnaire and structured likert scale.

ELIGIBILITY:
Inclusion Criteria:

* Adults who were able to understand Hindi and English.
* Who were willing to participate in the study.

Exclusion Criteria:

* Adults who were not available at the time of data collection.
* Adults having any psychological impairment.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of the present study was Adults residing in rural and urban area of Haryana.
  Target population:- Adults residing in rural areas and urban areas of Ambala District Haryana.
  Accessible population:- Adults residing in rural area (Mullana) and urban area (muncipal corporator ward number 14 and ward number 15 of Mahesh Nagar) of Ambala District Haryana and available during data collection.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Structured Questionnaire | 25-30 minutes
  One time assessment of knowledge of adults regarding adoption. Total score is calculated by finding the sum of the correct answer. Each correct answer scored as 1 and each incorrect answer scored as 0. It consists scale of scores 23-30 = Very Good, 19-22 = Good, 15-18 = Average, 0-14 = Below Average

SECONDARY OUTCOMES:
Likert Scale | 18-20 minutes
  3 point Likert Scale was used to assess opinion of adults regarding adoption. Total score is calculated by finding the sum of the 30 items. it consist 15 positive statements and 15 negative statements. Each positive statement scored as 3= agree, 2= uncertain,1=disagree and each negative statement scored as 3=disagree, 2=uncertain, 1= agree. it consists the scale of scores 68-90:Favourable 45-67: Moderately Favourable, 30-44: Unfavourable

CONTACTS AND LOCATIONS:
Overall Officials: Poonam Sheoran, Ph.D Nursing, Study Director — Maharishi Markandeshwar University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ezugwu FO, Obi SN, Onah HE. The knowledge, attitude and practice of child adoption among infertile Nigerian women. J Obstet Gynaecol. 2002 Mar;22(2):211-6. doi: 10.1080/01443610120113463. PMID 12521712